CLINICAL TRIAL: NCT01596140
Title: A Phase I Dose-Escalation Study of the BRAF Inhibitor Vemurafenib (Zelboraf®) in Combination With an mTOR Inhibitor, Everolimus (Afinitor®) or Temsirolimus (Torisel®), in Subjects With Advanced Cancer
Brief Title: Vemurafenib in Combination With Everolimus or Temsirolimus With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-0153; NCI-2012-00789 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2012-05-08; First posted 2012-05-10 (Estimated); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Advanced Cancer; Solid Tumor
Keywords: Vemurafenib; Everolimus; Afinitor; RAD001; temsirolimus; BRAF gene mutation; solid tumor; relapsed BRAF mutation positive malignant melanoma; refractory BRAF mutation positive malignant melanoma
MeSH Terms: interventions — Vemurafenib; Everolimus; temsirolimus; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Vemurafenib + Oral Everolimus (Experimental): Vemurafenib starting dose 720 mg orally twice day (morning/evening) for 28-day cycle plus Oral Everolimus starting dose 5 mg daily.
  Interventions: Drug: Vemurafenib; Drug: Everolimus
- Vemurafenib + Intravenous Temsirolimus (Experimental): Vemurafenib starting dose 720 mg orally twice day (morning/evening) for 28-day cycle plus Intravenous Temsirolimus starting dose 15 mg daily on Days 1, 8, 15, and 22 of each cycle.
  Interventions: Drug: Vemurafenib; Drug: Temsirolimus

INTERVENTIONS:
Drug: Vemurafenib — Starting dose 720 mg by mouth twice a day (3 tablets in the morning and 3 tablets in the evening) for 28-day study cycle.
  Other Names: Zelboraf®; PLX4032; RO5185426
Drug: Everolimus — Starting dose 5.0 mg by mouth daily for 28-day study cycle.
  Other Names: Afinitor®; RAD001
  Arms: Vemurafenib + Oral Everolimus
Drug: Temsirolimus — Starting dose 15 mg daily over 30-60 minutes on Days 1, 8, 15, and 22 of each 28-day cycle.
  Other Names: Temodar
  Arms: Vemurafenib + Intravenous Temsirolimus

SUMMARY:
The goal of this clinical research study is to find the highest tolerable dose of vemurafenib that can be given in combination with either everolimus or temsirolimus. The safety of these drug combinations will also be studied.

Vemurafenib is designed to block BRAF inside the cancer cells, which is a mutation that is involved in cancer cell growth.

Temsirolimus and everolimus are designed to block the growth of cancer cells, which may cause cancer cells to die.

DETAILED DESCRIPTION:
Study Drug Administration:

If you are found to be eligible to take part in this study, your doctor will decide whether you will receive either everolimus or temsirolimus

You will be assigned to a dose level of vemurafenib based on when you join this study. Up to 5 dose levels of vemurafenib will be tested. Up to 6 participants will be enrolled at each dose level. The first group of participants will receive the lowest dose level. Each new group will receive a higher dose than the group before it, if no intolerable side effects were seen. This will continue until the highest tolerable dose of vemurafenib is found.

Study Drug Administration:

You will take 3 vemurafenib tablets in the morning and 3 tablets in the evening.You will take it every day during each 28-day study cycle. You will take vemurafenib in combination with either 1 tablet of everolimus every day of each cycle or you will receive temsirolimus by vein over 30-60 minutes on Days 1, 8, 15, and 22 of each cycle.

You will receive a dosing diary to record ONLY the date and times when you did NOT take a scheduled dose of the study drug. You should bring this diary and any used or unused study drug bottles to your next study visit (even empty bottles must be returned).

Study Visits:

At all study visits, you will be asked about any drugs you may be taking and if you have had any side effects from them.

On Days 1 and 15 of Cycle 1 and Day 1 of Cycle 6:

* You will have a physical exam, including measurement of your vital signs.
* Your performance status will be recorded.
* Blood (about 3 teaspoons) will be drawn for routine tests.
* You will have an ECG (Day 15 only)

On Day 1 of Cycles 2 and 5:

* You will have a physical exam, including measurement of your vital signs.
* Your performance status will be recorded.
* Blood (about 3 teaspoons) will be drawn for routine tests.
* You will have an ECG.
* Your skin will be checked.
* You will have a CT scan or MRI scan to check the status of the disease (Cycle 5 only).

On Day 1 of Cycle 3:

* You will have a physical exam, including measurement of your vital signs.
* Your performance status will be recorded.
* Blood (about 3 teaspoons) will be drawn for routine tests.
* You will have an ECG.
* You will have a CT scan or MRI scan to check the status of the disease.

On Day 1 of Cycle 4:

* You will have a physical exam, including measurement of your vital signs.
* Your performance status will be recorded.
* Blood (about 3 teaspoons) will be drawn for routine tests.
* You will have an ECG.
* You will have a head and neck exam to check the status of the disease.

On Day 1 of Cycle 7:

* You will have a physical exam, including measurement of your vital signs.
* Your performance status will be recorded.
* Blood (about 3 teaspoons) will be drawn for routine tests.
* You will have a CT scan or MRI scan to check the status of the disease.
* You will have a head and neck exam to check the status of the disease.

On Day 1 of Cycles 8 and beyond:

* You will have a physical exam, including measurement of your vital signs.
* Your performance status will be recorded.
* Blood (about 3 teaspoons) will be drawn for routine tests.

After Cycle 7, every 12 weeks:

* You will have an ECG.
* You will have a head and neck exam to check the status of the disease.
* Your skin will be checked.

On Day 1 of every 2 cycles:

°You will have a CT scan or MRI scan to check the status of the disease.

Length of Study:

You may continue taking the study drugs for as long as the doctor thinks it is in your best interest. You will no longer be able to take the study drugs if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

Your participation on the study will be over once you have completed the follow-up.

End of Study Drug Dosing Visit:

Once you are no longer taking the study drug, you will have a study visit. At this visit:

* You will be asked about any drugs you may be taking and if you have had any side effects from them.
* You will have a physical exam, including measurement of your vital signs.
* Your performance status will be recorded.
* Blood (about 3 teaspoons) will be drawn for routine tests.
* You will have an ECG.
* You will have a CT scan or MRI scan to check the status of the disease.
* Your skin will be checked.

Safety Follow-Up Visit:

If you leave the study for any reason other than the disease getting worse, you will have a follow-up visit about 28 days after your last dose. At this visit:

* You will be asked about any drugs you may be taking and if you have had any side effects from them.
* You will have an ECG.
* Your skin will be checked.
* You will have a head and neck exam to check the status of the disease.

Follow-Up:

Every 3 months after the last dose of study drug (for up to 12 months) you will be contacted by phone and asked about any new drugs you may be taking. This should take less than 5 minutes. This follow up may be during a regularly scheduled clinic visit.

Participant Responsibilities:

* Take the study drug as instructed by the study staff.
* Keep your study appointments. If you cannot keep an appointment, reschedule as soon as you know that you will miss the appointment.
* Tell your doctor or study staff about any side effects, doctor visits, or hospitalizations that you may have.
* Keep the study drug in a safe place, for your use only, and away from children. It must be stored at room temperature but not warmer than 77 degrees F (25 degrees Celsius).
* Complete your diaries as instructed
* While on this study, you cannot take part in any other research project without approval from your doctor.

This is an investigational study. Vemurafenib is FDA-approved for metastatic melanoma. Its use in other types of cancer is investigational. Everolimus and temsirolimus are FDA approved kidney cancer. The combination of these drugs is investigational.

Up to 114 participants will be enrolled in this study. All will take part at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmation of BRAF mutation-positive malignancy is required for selection of patients for vemurafenib therapy
2. Measurable or non-measurable disease by RECIST 1.1.
3. Patients with advanced cancer should be refractory to standard therapy, relapsed after standard therapy, or have no standard therapy available that improves survival by at least three months.
4. Patients must be at least 3 weeks past receiving cytotoxic therapy and at least 5 half-lives after their previous treatment or 3 weeks, whichever is shorter, after biologic therapy. Patients may receive palliative radiotherapy immediately or during treatment provided that not all target lesions are radiated.
5. ECOG performance status </= 2 (Karnofsky >/= 60%; Lansky Score >/= 50).
6. Patients must have normal organ and marrow function defined as: absolute neutrophil count >/=1,000/mL; platelets >/=50,000/mL; creatinine < 2.0; total bilirubin < 2.0; ALT(SGPT) </= 3 X ULN; Exception for patients with liver metastasis: ALT(SGPT) </= 5 X ULN.
7. Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 30 days after the last dose.
8. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Patients with uncontrolled concurrent illness, including but not limited to: ongoing or active infection requiring hospitalization; psychiatric illness/social situations that would limit compliance with study requirements.
2. Exclusion of patients with creatinine >2.0 and bilirubin > 2.0.
3. Pregnant or lactating women.
4. Patients with a history of bone marrow transplant within the previous two years.
5. Patients with a known hypersensitivity to any of the components of the drug products.
6. Patients with major surgery within 30 days prior to entering the study.
7. Patients with a baseline QTc > 500 ms.
8. Patients who are unable to swallow pills.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2012-12-18 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of Combination Vemurafenib | First cycle of 28 day cycle
  The MTD of combination Vemurafenib and Everolimus or Vemurafenib and Temsirolimus is defined as the highest dose studied in which the incidence of dose limiting toxicity (DLT) was less than one third (33%) of the participants at that dose level. DLT defined as any Grade 3 or 4 non-hematologic toxicity, as defined in NCI CTC v4.0, even if expected and believed related to study medications, any Grade 4 hematologic toxicity lasting two weeks or longer despite supportive care; Grade 3 nausea/vomiting > 48 hours or any Grade 4 nausea/vomiting; and any other Grade 3 non-hematologic toxicity, including symptoms/signs of vascular leak or cytokine release syndrome; or any severe or life-threatening complication or abnormality not defined in NCI-CTCAE that is attributable to therapy.

SECONDARY OUTCOMES:
Tumor Response | 4 months
  Tumor response defined as one or more of the following: (1) stable disease for more than or equal to 4 months, (2) decrease in measurable tumor (sentinel lesions) by more than or equal to 20% by RECIST criteria, (3) decrease in tumor markers by more than or equal to 25% (for example, a >/= 25% decrease in CA125 for patients with ovarian cancer), or (4) a partial response according to Choi criteria, i.e., decrease in size by 10% or more, or a decrease in tumor density, as measured in Hounsfield units (HU), by more than or equal to 15%.

CONTACTS AND LOCATIONS:
Overall Officials: Vivek Subbiah, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org